CLINICAL TRIAL: NCT06184594
Title: Developing and Testing a Digital Toolkit to Improve Colorectal Cancer Screening Rates in Federally Qualified Health Centers
Brief Title: Evaluating the Efficacy of the eNav Toolkit to Improve Colorectal Cancer Screening
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: The Institute for Family Health (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sarah Miller, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY-20-01888; R01CA248981 (NIH)
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer Screening
Keywords: Colorectal Cancer; Screening; Federally Qualified Health Centers; Digital Patient Navigation Toolkit
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eNav intervention (Experimental): Subjects assigned to this arm will receive a link to the eNav website.
  Interventions: Other: eNav
- Usual Care Group (Placebo Comparator): Subjects assigned to this arm will not receive the link to the website and will receive standard clinical care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: eNav — The eNav toolkit is a digital navigation toolkit that includes a website and text messaging support. The website includes information, motivational support, decisional support and cues to action (e.g., ability to request a CRC screening test). The eNav tool also includes text-messaging based navigation (e.g., reminders, instructions to complete the screening test).
  Arms: eNav intervention
Other: Standard of Care — Standard of care procedures for selecting their CRC screening test.
  Arms: Usual Care Group

SUMMARY:
The purpose of this research study is to evaluate the efficacy of a digital navigation tool, called the eNav to improve colorectal cancer screening uptake among patients treated at federally qualified health centers (FQHC)s. The digital navigation tool includes a website and text messaging support. The website includes information, motivational support, decisional support and cues to action (e.g., ability to request a CRC screening test). The eNav tool also includes text-messaging based navigation (e.g., reminders, instructions to complete the screening test).

DETAILED DESCRIPTION:
This is a multi-site randomized clinical trial to evaluate the efficacy of the eNav Toolkit. A total of 400 participants will be from four FQHC clinics within the Institute for Family Health FQHC network. Participants will be randomly assigned to one of two groups:

1. eNav group (N=200) or
2. usual care group (N=200)

Participants will consent and complete a baseline questionnaire (demographics, medical information) 1-4 weeks before their primary care appointment.

Those in the intervention group will receive a link to the eNav website. The digital navigation tool includes a website and text-messaging support. The website includes information, motivational support, decisional support and cues to action (e.g., ability to request a CRC screening test). The eNav tool also includes text-messaging based navigation (e.g., reminders, instructions to complete the screening test).

The control group will receive standard clinical care.

Then 3-6 weeks after that primary care appointment, the research team will reach out to participants to complete a follow-up questionnaire. The follow up questionnaire will assess constructs guided by the health belief model (e.g., self-efficacy, benefits/barriers for CRC screening).

The impact of the eNav Toolkit on CRC screening completion at 6 months will be evaluated by checking their medical records. If a patient does not have a CRC screening recorded in their medical record, the research team will call the patient to inquire whether they have completed the CRC screening.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated at the Institute for Family Health (IFH)
* Patient 45 to 75 years old
* English or Spanish speaking
* Able to provide consent within the study time frame (within a month of the primary care appointment
* Patients have access to a computer, tablet or mobile device to access the eNav Toolkit OR willing to use a clinic provided device, in person at either IFH OR Mount Sinai
* Patient scheduled for a primary care appointment at IFH
* Patients are due for colorectal cancer screening (as determined by the health maintenance alert in the medical chart)

Exclusion Criteria:

* Unable to provide informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Colorectal Cancer (CRC) Screening completion | End of study, at 6 months
  CRC, Yes/No
  Medical chart review will determine whether the CRC screening was complete. If a patient does not have a CRC screening result recorded in their medical record, the research team will call the patient to inquire whether they have completed the CRC screening.

SECONDARY OUTCOMES:
Number of participants who complete screening tests with adequate quality | End of study, at 6 months
  The number of participants who complete the screening test (i.e., colonoscopy, FIT or FIT-DNA) with adequate quality. Test quality will be coded as "inadequate" if the test needs to be repeated or cannot be resulted due to inadequate quality (e.g., poor bowel prep, inadequate stool sample).
Number of participants who complete the screening test with inadequate preparation | End of study, at 6 months
  The number of participants who complete the screening test and the preparation is inadequate (e.g., poor bowel prep quality, inadequate stool sample collection).
Adherence to follow up recommendations | End of study, at 6 months
  Record if the study participant is following the colorectal cancer screening recommendations after the CRC test has been completed. Measured as:
  Yes = participant completed the recommended follow up No = participant did NOT complete the recommended follow up In process = the recommended follow up does not fall within the 6-month time frame Missing = data not available in the medical chart
The Colorectal Cancer Screening Beliefs Instrument Score | Approximately 3-4 weeks after primary care appointment
  The assessments specifically measure the following Health Belief Model scales:
  * Perceived Benefits of Stool-based Tests: min 3 - max 15
  * Perceived Benefits of Colonoscopy: min 3 - max 15
  * Perceived Susceptibility: min 2 - max 10
  * Perceived Barriers of Stool-Based Tests: min 7 - max 35
  * Perceived Barriers of Colonoscopy: min 9 - max 45
  * Perceived Self-Efficacy of Stool-based Tests: min 8 - max 40
  * Perceived Self-Efficacy of Colonoscopy: min 12 - max 60
  * Perceive Severity: min 3 - max 15
  Higher scores indicate greater benefit/barriers levels of the scale (e.g., higher scores = more barriers, more benefits, higher perceived susceptibility of CRC, higher levels of self-efficacy), there is no summed score.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Miller, PsyD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.